CLINICAL TRIAL: NCT05423795
Title: A Multifaceted Telemedicine-Based Intervention to Improve Outcomes of Cancer Patients Admitted to the ICU : A Stepped Wedge Cluster-randomised Trial
Brief Title: A Multifaceted Telemedicine-Based Intervention to Improve Outcomes of Cancer Patients Admitted to the ICU
Acronym: EXPERT-IS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: P 150954J
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Active Malignancies; Life Threatening Complication of the Malignancy or Its Treatments

STUDY DESIGN:
Intervention Model Description: Stepped wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator Arm (Other): Classic expertise (as routinely performed in the participating ICU)
  Interventions: Other: Standard of care arm
- Telemedicine-based intervention (Experimental): Telemedicine-based expert advice.
  Interventions: Other: Telemedicine-based intervention

INTERVENTIONS:
Other: Telemedicine-based intervention — Telemedicine-based intervention Multifaceted intervention including daily videoconferences with audit and feedback, educational interventions, and dissemination of published works
  Arms: Telemedicine-based intervention
Other: Standard of care arm — Classic expertise (as routinely performed in the participating ICU)
  Arms: Comparator Arm

SUMMARY:
Admission to the intensive care unit (ICU) is a common event in patients treated for solid tumors or hematologic malignancies. A volume-outcome relationship has been shown in these patients, with a mortality rate decreasing from 70% in low-volume centres to 30-40% in high-volume centres.

We hypothesize that providing the low-volume centres with assistance from experts working in high-volume centres for the management of critically-ill cancer patients can bring down mortality to the values seen in high-volume centres.

The main objective of this study is to evaluate whether combining three knowledge-transfer methods (videoconference-based forum, educational sessions, and dissemination of published work) increases the survival of cancer patients managed in low-volume centres to the values seen in high-volume centres.

The main endpoint is all-cause mortality at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (> 18 years old)
2. Active malignancy;
3. ICUs seeking for an advice must admit fewer than 30 patients with active cancer per year;
4. Patients has been urgently admitted in the ICU for a life threatening complication of the malignancy or its treatments.

Exclusion Criteria:

1. Isolated HIV infection or AIDS;
2. ICU admission complicating scheduled surgery,
3. Treatment-limitation decisions at admission;
4. No coverage by the French statutory health insurance system,
5. Pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | at hospital discharge (up to 28 days)

SECONDARY OUTCOMES:
Number of changes based on expert opinion | at 28 days
Number of invasive diagnostic tests used | at 28 days
Number of non-invasive diagnostic tests used | at 28 days
Proportion of patients with non-invasive ventilation and/or high flow oxygen | at 28 days
Proportion of patients in whom the cause for ICU admission remained undetermined | at 28 days
Number of days without life-supporting interventions | at 28 days
Number of anti-microbial agents | at 28 days
Number of blood transfusions | at 28 days
Number of chemotherapy | at 28 days
Proportion of patients with antibiotic de-escalation | at 28 days
Duration of antibiotic therapy | up to 28 days
Length of ICU stay | at hospital discharge (up to 28 days)
Proportion of ICU-acquired events | at 28 days
Satisfaction of patients, intensivists, primary physicians, and expert. | at 28 days
  Satisfaction will be assessed using a visual analog scale (VAS). The VAS is a scale ranging from 0 to 10, with a higher score indicating greater satisfaction.

IPD SHARING:
Plan to Share IPD: Undecided